CLINICAL TRIAL: NCT06214533
Title: Celiac Plexus Block to Reduce Opioid Consumption Following Hepato-pancreato-biliary Mini-invasive Surgery: a Randomized Controlled Trial
Brief Title: Celiac plExus Block to Reduce OpioID Consumption Following Hepato-pancreato-biliary Mini-invasive Surgery
Acronym: CEBOIDS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022-090
Record Dates: First submitted 2023-04-03; First posted 2024-01-19 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Pancreatic Ductal Adenocarcinoma; Liver, Cancer of, Primary Resectable
Keywords: laparoscopic hepato-pancreato-biliary surgery
MeSH Terms: interventions — Ropivacaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Never block (Experimental): Prior to the end of the laparoscopic surgery and any additional procedures, the bilateral celiac plexus block will be performed by the surgeon after identification of the aorta at the superior border of body of pancreas. A 22-gauge spinal needle will be inserted into the retroperitoneal fat on either side of the aorta under direct vision. Needle aspiration will be performed to exclude entry into vessels before administration of the interventional drug.
  The block will contain 20 mL of 0.5% ropivacaine hydrochloride + 1:400000 adrenaline.
  Intervention: Drug: 20 mL of 0.5% Ropivacaine
  Interventions: Drug: Ropivacaine 0.5%
- Placebo block (Placebo Comparator): Patients in the control arm will undergo the celiac plexus block procedure as well. The block will contain 20 ml of 0.9% normal saline + 1:400000 adrenaline.
  Intervention: Drug: 20 mL of 0.9% normal saline
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Ropivacaine 0.5% — Prior to the end of the laparoscopic surgery and any additional procedures, the bilateral celiac plexus block will be performed by the surgeon after identification of the aorta at the superior border of body of pancreas. A 22-gauge spinal needle will be inserted into the retroperitoneal fat on either side of the aorta under direct vision. Needle aspiration will be performed to exclude entry into vessels before administration of the interventional drug. The block will contain 20 mL of 0.5% ropivacaine hydrochloride + 1:400000 adrenaline.
  Other Names: Naropin
  Arms: Never block
Drug: Normal Saline — Prior to the end of the laparoscopic surgery and any additional procedures, the bilateral celiac plexus block will be performed by the surgeon after identification of the aorta at the superior border of body of pancreas. A 22-gauge spinal needle will be inserted into the retroperitoneal fat on either side of the aorta under direct vision. Needle aspiration will be performed to exclude entry into vessels before administration of the interventional drug. The block will contain 20 ml of 0.9% normal saline + 1:400000 adrenaline.
  Arms: Placebo block

SUMMARY:
The goal of this study is to assess the efficacy of intraoperative celiac plexus block (CPB) to reduce opioid consumption following laparoscopic hepato-pancreato-biliary surgery

DETAILED DESCRIPTION:
A bilateral CPB is convenient and safe to perform under the direct laparoscopic vision of the surgeons during surgery; however, perspective data are warranted. The investigators hypothesize that a bilateral CPB using 0.5% ropivacaine will improve the quality of recovery following a laparoscopic hepato-pancreato-biliary surgery. The primary endpoint is the Postoperative opioid use. Secondary endpoints include acute postoperative pain, opioid consumption, the incidence of postoperative nausea or vomiting (PONV), the 15-item quality of recovery questionnaire (QoR-15), length of post-anesthesia care unit (PACU) stay, length of post-operative hospital stay, and chronic post-surgical pain at 90 d after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Over age 18
* Undergoing laparoscopic hepato-pancreato-biliary surgery

Exclusion Criteria:

* Patient refuse
* Relatively contraindications: severe heart, liver, or kidney dysfunction, coagulation dysfunction, and local anesthetic allergy history
* Intervention unlikely to be effective: drug abuse history, receiving other types of nerve block treatment
* Unlikely to complete the follow-up: alcoholism, planned to replace WeChat and phone within three months; the expected life span less than three months
* Unable to cooperate with the questionnaire and use the patient-controlled analgesia pump

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative opioid use | Up to 24 h after surgery
  The primary outcome will be morphine equivalent during the first postoperative 24 h

SECONDARY OUTCOMES:
Postoperative opioid use | Up to 72 h after surgery
  Patients will be recorded for up to 72 h postoperative opioid consumption.
Numeric rating scale (NRS) for pain | Up to 72 h after surgery
  Patients will be asked to complete a daily diary up to 72 h that records numeric pain rating scale
Postoperative vomiting | Up to 72 h after surgery
  Incidence of postoeprative vomiting will be recorded for up to 72 h
Quality of recovery using the 15-item quality of recovery questionnaire (QoR-15) | Up to 72 h after surgery
  Patients will be asked to complete a 15-item quality of recovery questionnaire up to 72 h after surgery
Post-anesthesia care unit (PACU) time | Through study completion, an average of 1 year
  Length of PACU stay
Post-operative hospital time | Through study completion, an average of 1 year
  Length of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Ruan, Principal Investigator — The Sixth Affiliated Hospital, Sun Yat-sen University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sommer M, de Rijke JM, van Kleef M, Kessels AG, Peters ML, Geurts JW, Gramke HF, Marcus MA. The prevalence of postoperative pain in a sample of 1490 surgical inpatients. Eur J Anaesthesiol. 2008 Apr;25(4):267-74. doi: 10.1017/S0265021507003031. Epub 2007 Dec 6. PMID 18053314
- [Background] Poon RT, Fan ST, Lo CM, Ng IO, Liu CL, Lam CM, Wong J. Improving survival results after resection of hepatocellular carcinoma: a prospective study of 377 patients over 10 years. Ann Surg. 2001 Jul;234(1):63-70. doi: 10.1097/00000658-200107000-00010. PMID 11420484
- [Background] Al Samaraee A, Rhind G, Saleh U, Bhattacharya V. Factors contributing to poor post-operative abdominal pain management in adult patients: a review. Surgeon. 2010 Jun;8(3):151-8. doi: 10.1016/j.surge.2009.10.039. Epub 2010 Feb 12. PMID 20400025
- [Background] Kehlet H. Multimodal approach to control postoperative pathophysiology and rehabilitation. Br J Anaesth. 1997 May;78(5):606-17. doi: 10.1093/bja/78.5.606. PMID 9175983
- [Background] McLeod RS, Aarts MA, Chung F, Eskicioglu C, Forbes SS, Conn LG, McCluskey S, McKenzie M, Morningstar B, Nadler A, Okrainec A, Pearsall EA, Sawyer J, Siddique N, Wood T. Development of an Enhanced Recovery After Surgery Guideline and Implementation Strategy Based on the Knowledge-to-action Cycle. Ann Surg. 2015 Dec;262(6):1016-25. doi: 10.1097/SLA.0000000000001067. PMID 25692358
- [Background] Ladha KS, Patorno E, Huybrechts KF, Liu J, Rathmell JP, Bateman BT. Variations in the Use of Perioperative Multimodal Analgesic Therapy. Anesthesiology. 2016 Apr;124(4):837-45. doi: 10.1097/ALN.0000000000001034. PMID 26835644
- [Background] Gan TJ. Poorly controlled postoperative pain: prevalence, consequences, and prevention. J Pain Res. 2017 Sep 25;10:2287-2298. doi: 10.2147/JPR.S144066. eCollection 2017. PMID 29026331
- [Background] Tan M, Law LS, Gan TJ. Optimizing pain management to facilitate Enhanced Recovery After Surgery pathways. Can J Anaesth. 2015 Feb;62(2):203-18. doi: 10.1007/s12630-014-0275-x. Epub 2014 Dec 10. PMID 25501696
- [Background] Revie EJ, Massie LJ, McNally SJ, McKeown DW, Garden OJ, Wigmore SJ. Effectiveness of epidural analgesia following open liver resection. HPB (Oxford). 2011 Mar;13(3):206-11. doi: 10.1111/j.1477-2574.2010.00274.x. PMID 21309939
- [Background] Tzimas P, Prout J, Papadopoulos G, Mallett SV. Epidural anaesthesia and analgesia for liver resection. Anaesthesia. 2013 Jun;68(6):628-35. doi: 10.1111/anae.12191. PMID 23662750
- [Background] Teo ZHT, Tey BLJ, Foo CW, Wong WY, Low JK. Intraoperative Celiac Plexus Block With Preperitoneal Infusion Reduces Opioid Usage in Major Hepato-pancreato-biliary Surgery: A Pilot Study. Ann Surg. 2021 Jul 1;274(1):e97-e99. doi: 10.1097/SLA.0000000000004883. PMID 33856374
- [Background] Kambadakone A, Thabet A, Gervais DA, Mueller PR, Arellano RS. CT-guided celiac plexus neurolysis: a review of anatomy, indications, technique, and tips for successful treatment. Radiographics. 2011 Oct;31(6):1599-621. doi: 10.1148/rg.316115526. PMID 21997984
- [Background] Zhu J, Jin Z. Interventional Therapy for Pancreatic Cancer. Gastrointest Tumors. 2016 Oct;3(2):81-89. doi: 10.1159/000446800. Epub 2016 Sep 6. PMID 27904860
- [Background] Penman ID. Coeliac plexus neurolysis. Best Pract Res Clin Gastroenterol. 2009;23(5):761-6. doi: 10.1016/j.bpg.2009.05.003. PMID 19744638
- [Background] Lavu H, Lengel HB, Sell NM, Baiocco JA, Kennedy EP, Yeo TP, Burrell SA, Winter JM, Hegarty S, Leiby BE, Yeo CJ. A prospective, randomized, double-blind, placebo controlled trial on the efficacy of ethanol celiac plexus neurolysis in patients with operable pancreatic and periampullary adenocarcinoma. J Am Coll Surg. 2015 Apr;220(4):497-508. doi: 10.1016/j.jamcollsurg.2014.12.013. Epub 2014 Dec 17. PMID 25667135
- [Background] Liu S, Fu W, Liu Z, Liu M, Ren R, Zhai H, Li C. MRI-guided celiac plexus neurolysis for pancreatic cancer pain: Efficacy and safety. J Magn Reson Imaging. 2016 Oct;44(4):923-8. doi: 10.1002/jmri.25246. Epub 2016 Mar 28. PMID 27019192
- [Background] Wyse JM, Carone M, Paquin SC, Usatii M, Sahai AV. Randomized, double-blind, controlled trial of early endoscopic ultrasound-guided celiac plexus neurolysis to prevent pain progression in patients with newly diagnosed, painful, inoperable pancreatic cancer. J Clin Oncol. 2011 Sep 10;29(26):3541-6. doi: 10.1200/JCO.2010.32.2750. Epub 2011 Aug 15. PMID 21844506
- [Background] Sakorafas GH, Tsiotou AG, Sarr MG. Intraoperative celiac plexus block in the surgical palliation for unresectable pancreatic cancer. Eur J Surg Oncol. 1999 Aug;25(4):427-31. doi: 10.1053/ejso.1999.0670. No abstract available. PMID 10419716
- [Background] Kretzschmar M, Krause J, Palutke I, Schirrmeister W, Schramm H. [Intraoperative neurolysis of the celiac plexus in patients with unresectable pancreatic cancer]. Zentralbl Chir. 2003 May;128(5):419-23. doi: 10.1055/s-2003-40039. German. PMID 12813642
- [Background] Lillemoe KD, Cameron JL, Kaufman HS, Yeo CJ, Pitt HA, Sauter PK. Chemical splanchnicectomy in patients with unresectable pancreatic cancer. A prospective randomized trial. Ann Surg. 1993 May;217(5):447-55; discussion 456-7. doi: 10.1097/00000658-199305010-00004. PMID 7683868
- [Background] Strong VE, Dalal KM, Malhotra VT, Cubert KH, Coit D, Fong Y, Allen PJ. Initial report of laparoscopic celiac plexus block for pain relief in patients with unresectable pancreatic cancer. J Am Coll Surg. 2006 Jul;203(1):129-31. doi: 10.1016/j.jamcollsurg.2006.03.020. Epub 2006 May 30. No abstract available. PMID 16798497
- [Background] Allen PJ, Chou J, Janakos M, Strong VE, Coit DG, Brennan MF. Prospective evaluation of laparoscopic celiac plexus block in patients with unresectable pancreatic adenocarcinoma. Ann Surg Oncol. 2011 Mar;18(3):636-41. doi: 10.1245/s10434-010-1372-x. Epub 2010 Oct 17. PMID 20953910